CLINICAL TRIAL: NCT01540084
Title: Cocktail Sedation Containing Propofol Versus Conventional Sedation for ERCP: a Prospective, Randomized Controlled Study
Brief Title: Cocktail Sedation Containing Propofol Versus Conventional Sedation for Endoscopic Retrograde Cholangiopancreatography (ERCP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, MD, Principal investigator, King Chulalongkorn Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PA-001
Record Dates: First submitted 2012-02-16; First posted 2012-02-28 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Disorders of Gallbladder, Biliary Tract and Pancreas
Keywords: Cocktail sedation; ERCP
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional group (Active Comparator): For induction, 25 mg of meperidine and 2.5 mg of midazolam were administered. To maintain conscious level of patient at moderate or deep level, 25 mg of meperidine and/or 2.5 mg of midazolam were administered as necessary.
  Interventions: Drug: propofol
- cocktail group (Experimental): For induction, 25 mg of meperidine and 2.5 mg of midazolam were administered. To maintain conscious level of patient at moderate or deep level, 1% propofol at the rate of 1 mg/kg/hr was administered. An additional 0.5 mg/kg bolus was administered as needed to achieve the designed conscious level.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — For induction, 25 mg of meperidine and 2.5 mg of midazolam were administered in both groups. In the cocktail group, one milligram per kilogram body weight of 1% propofol emulsion (Baxter Healthcare Corp., Irvine, CA) was slowly infused by an automated pump (Terufusion syringe pump TE-331, Terumo Corporation, Tokyo, Japan). To maintain conscious level of patient in the conventional group to be at moderate or deep level, 25 mg of meperidine and/or 2.5 mg of midazolam were administered as necessary, whereas patients in the cocktail group were continuously administered with 1% propofol at the rate of 1 mg/kg/hr. An additional 0.5 mg/kg bolus was administered as needed to achieve the designed conscious level.
  Other Names: diprivan

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) practically requires moderate to deep sedation by a combination of benzodiazepine and opioid. Propofol as a sole agent may cause oversedation. A combination (cocktail) of infused propofol, meperidine, and midazolam can reduce the dosage of propofol and may result in a lower risk of oversedation. The investigators prospectively compare the efficacy, recovery time, patient satisfactory, and side effects between cocktail and conventional sedations in patients undergoing ERCP.

DETAILED DESCRIPTION:
ERCP patients were prospectively randomized into 2 groups; the cocktail group and the controls. For induction, a combination of 25 mg of meperidine and 2.5 mg of midazolam were injected in both groups. In the cocktail group, a bolus dose of propofol 1 mg/kg was administered and continuously infused. In the controls, 25 mg of meperidine or 2.5 mg/kg of midazolam were titrated to maintain the level of sedation.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for ERCP

Exclusion Criteria:

* Age under 18 years
* American Society of Anesthesiologists' (ASA) physical classification IV - V
* History of sulfite, egg or soy bean allergy
* Emergency need for ERCP
* Informed consent could not be obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2006-12; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
procedure related time | participants will be followed for the duration of procedure, an expected average of 1.5 hours
  (1) induction time (the time from sedation to scope intubation), (2) procedural time (the time from scope intubation to scope withdrawal), and (3) recovery time (the time from scope withdrawal to full recovery (modified Aldrete score of 10)). The induction time and procedural time were recorded by the nurse in the endoscopy unit.

SECONDARY OUTCOMES:
Cardiopulmonary complications | participants will be followed for the duration of procedure, an expected average of 1.5 hours
  (1) hypotension (systolic blood pressure drops to less than 90 mmHg or decreases more than 25% from the baseline), (2) bradycardia (heart rate <40 beats/min), (3) desaturation (oxygen saturation <90% for >10 seconds), and (4) apnea (cessation of respiratory activity for over 10 seconds under visual observation). If the oxygen saturation dropped to <85% for more than 30 seconds despite oxygen supplementation or apnea occurred, the procedure would be interrupted and reversal medications would be given to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Rungsun Rerknimitr, MD, Principal Investigator — Gastroenterology unit, King Chulalongkorn Memorial Hospital
Locations (1):
- Gastroenterology Unit, King Chulalongkorn Memorial Hospital, Patumwan, Bangkok, Thailand

REFERENCES:
- [Derived] Angsuwatcharakon P, Rerknimitr R, Ridtitid W, Kongkam P, Poonyathawon S, Ponauthai Y, Sumdin S, Kullavanijaya P. Cocktail sedation containing propofol versus conventional sedation for ERCP: a prospective, randomized controlled study. BMC Anesthesiol. 2012 Aug 9;12:20. doi: 10.1186/1471-2253-12-20. PMID 22873637